CLINICAL TRIAL: NCT04020796
Title: Acute Effects of Beet Juice Intake on Vascular Function in Treated Hypertensive Patients
Brief Title: Acute Effects of Beet Juice Intake on the Vascular Function of Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Pedro Ernesto (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Samanta De Souza Mattos, Nutritionist, Hospital Universitario Pedro Ernesto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: BRJ-700
Record Dates: First submitted 2019-06-28; First posted 2019-07-16 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: randomized, crossover, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot juice (Active Comparator): Randomized cross-over trial. Thirty-seven hypertension, age 40-70 years were randomized to receive a 500ml volume of beetroot juice in a single moment.
  Interventions: Dietary Supplement: Beetroot juice
- Mineral water (Placebo Comparator): Randomized cross-over trial. Thirty-seven hypertension, age 40-70 years were randomized to receive a 500ml volume of mineral water in a single moment.
  Interventions: Dietary Supplement: Beetroot juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice — Thirty-seven hypertension, with age 40-70 years were randomized to receive a 500ml volume of beetroot juice contains 11.5 mmol of inorganic nitrate or mineral water in a single moment.

SUMMARY:
To assess the acute effects of only one dose of beet juice on hypertensive subjects treated with vascular endothelial function parameters, using the microvascular reactivity method.

DETAILED DESCRIPTION:
Systemic arterial hypertension is an established risk factor for cardiovascular disease (CVD). Among the main modifiable environmental factors of hypertension, the investigators highlight inadequate eating habits, such as low vegetable consumption. Clinical studies have shown that inorganic nitrate from beet juice intake has a protective effect against CVD due to reduced blood pressure, inhibition of platelet aggregation and prevention of endothelial dysfunction. However, there is still no consensus on its benefits of inorganic nitrate in vascular health. Associated with this, there are no previous studies in the literature that correlate the acute effects of inorganic nitrate intake on endothelial function assessed by microvascular reactivity through laser. The objective of the present study is to evaluate the acute effects (single dose) of inorganic nitrate, through the ingestion of beet juice, in the vascular parameters and endothelial function of treated hypertensive patients of both sexes.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* Age between 40 and 70 years
* Previous diagnosis of primary systemic arterial hypertension
* Signed the Informed Consent Term.

Exclusion Criteria:

* Secondary hypertension
* Systolic blood pressure greater than or equal to 180 mmHg or diastolic BP greater than or equal to 110 mmHg
* In use of beta-blockers
* Diabetes mellitus
* History of cancer
* Use of any dietary supplement
* Any serious life-threatening illness
* Cardiovascular diseases

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Microvascular reactivity | 150 minutes
  A laser speckle contrast imaging system with a laser wavelength of 785 nm system will measure non-invasively real time cutaneous microvascular flow changes in the forearm. For the post occlusive reactive hyperemia test, arterial occlusion will be performed with suprasystolic pressure (50 mmHg above the systolic arterial pressure) using a sphygmomanometer applied to the arm of the subject over three minutes. Peak skin flow will be measured after pressure release.

SECONDARY OUTCOMES:
Central blood pressure | 150 minutes
  Central systolic blood pressure, diastolic blood pressure, mean arterial pressure and pulse pressure before and after intervention and their potential effects on changes in subendocardial viability ratio and ejection duration after intervention with beetroot juice and water.

CONTACTS AND LOCATIONS:
Overall Officials: Samanta S Mattos, Principal Investigator — State University of Rio de Janeiro; Mario F Neves, MD, PhD, Study Director — State University of Rio de Janeiro
Locations (1):
- Samanta de Souza Mattos, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD with other researchers